CLINICAL TRIAL: NCT04020562
Title: Effects of a Mild Resistive Expiratory Technique on Pulmonary Functions of Spinal Cord Injury
Brief Title: Mild Resistive Expiratory Breathing Technique On Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Faiza Irshad
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries
Keywords: Pulmonary Function Test; Spinal Cord; Breathing Exercise; Expiratory
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild Resistive Expiratory Technique (Experimental): Mild resistive Expiratory Technique from EMST150- five-week training protocol.
  Interventions: Other: Mild Resistive Expiratory Technique
- Conventional Training (Active Comparator): Breathing exercise, Assistive Coughing, ROM Exercises, Sustained stretching, Splinting, Bracing, Functional Mobility, Tilt table standing
  Interventions: Other: Conventional Training

INTERVENTIONS:
Other: Mild Resistive Expiratory Technique — Mild Resistive Expiratory Technique (EMST150- five-week training protocol):
  The EMST requires the participant to forcibly blow into the device for 5 seconds with sufficient pressure to open the one-way valve. Each "blow" is one repetition. The device will be set at a resistance of 30 cmH2O. Participants will be instructed to complete five sets of five repetitions (total of 25 times and approximately 20 minutes per day), any five days per week, for five weeks. Whole exercise will be done in sitting position. Rest between repetitions will be given according to comfort level of patient.
  Arms: Mild Resistive Expiratory Technique
Other: Conventional Training — Breathing exercise: Deep breathing 10-15 repetitions twice a day. Assistive Coughing: 5-6 repetitions twice a day. ROM Exercises: Both active and passive limb ROM exercises 10-15 repetitions twice a day.
  Sustained stretching: Both upper and lower limbs, 10 repetitions, held for 5 seconds, twice a day.
  Splinting: According to patient's injury level Bracing: According to patient's injury level Functional Mobility: Mobilizing patient according to injury level Tilt table standing: 10-15 minutes once a day
  Arms: Conventional Training

SUMMARY:
Studies have been conducted on the effectiveness of inspiratory muscle training on tetraplegics, and less has been reported on expiratory muscle training on paraplegics; especially in Pakistan there was no such study done up-to my knowledge. Paraplegic individuals develop pulmonary complications due to prolonged general immobilization of body and ineffective cough due to respiratory muscle weakness. This study will identify the effects of expiratory muscle training using "Expiratory Muscle Strength Trainer- 150" in paraplegic individuals in Peshawar, Pakistan

DETAILED DESCRIPTION:
A study on the effects of accessory expiratory muscle training and showed that there was a significant improvement in vital capacity of experimental group. The investigator recruited 40 patients and randomly allocated them to control and experimental groups. Experimental group received expiratory muscle training for half hour a day, six days a week for eight weeks, which included training using PFLEX muscle trainer. Control group received conventional breathing exercises and assistance in coughing. Experimental group showed improvement in mean vital capacity from 1.48 to 1.98 liters and in mean expiratory muscle strength from 43.76 cmH2O to 68 cmH2O. Control group yielded no changes.

A respiratory muscle training and electrical stimulation of abdominal muscles on thirteen quadriplegic individuals to assess their respiratory function. The study consisted of training the patients for three months. Each subject was given one-month inspiratory training, followed by second month of expiratory muscle training, and then last month without training. Vital capacity showed 19% increase in the experimental group while control group showed no improvement .

A randomized controlled trial to assess the effect of expiratory muscle training on pulmonary function of 29 spinal cord injury patients in an acute inpatient rehabilitation hospital. Patients were randomized into two groups. Experimental group consisting of 16 patients received expiratory muscle training using EMST for 10 repetitions twice a day, 5 days a week, for 6 weeks. Control group consisted of 13 individuals and they received sham training. There was no significant difference reported between both groups

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury (level T1 and Below)
* Paraplegic

Exclusion Criteria:

* Rib fractures
* Active inflammation or infection going in body
* Diagnosed (primary Lung Diseases)
* Individuals with psychiatric disorders or malignancies

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow (PEF) | 5th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze peak expiratory flow PEF in Liter/second
Forced Expiratory Volume in 1 second (FEV1) | 5th week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced Expiratory Volume in 1 second FEV1 in Liters
Forced vital Capacity (FVC) | 5th Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze Forced vital Capacity in Liters
FEV1/ FVC Ratio | 5th Week
  Changes from the Baseline, the digital spirometer is used in clinical setting to analyze ratio between Forced Expiratory Volume in 1 second and Forced vital Capacity.

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS) | 5th week
  It is a 5-item scale designed to measure the global cognitive perceptions of an individual's life satisfaction. Participants indicate how much they agree or disagree with each of the 5 items in the questionnaire using a 7-point scale that ranges from 7 which corresponds to "strongly agree" to 1 which corresponds to "strongly disagree" . This scale shows good convergent validity with other scales and with other types of assessments of subjective well-being. SWLS shows high internal consistency and high temporal reliability. It has shown to have sufficient sensitivity to detect changes in life satisfaction during the period of clinical intervention. Changes from baseline
The Patient Health Questionnaire (PHQ-9) | 5th Week
  It is a 9-item self-administered questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression. It rates the frequency of symptoms. Each question has scale of answers from 0 which represents "not at all" to 3 which represents "nearly every day". The diagnostic validity of this questionnaire was assessed by using it on 6000 patients in 8 primary care clinics and 7 obstetrical clinics. A score of >10 on PHQ-9 had both sensitivity and specificity of 88% for major depression. PHQ-9 score of 5 represents mild, while 10, 15, and 20 represent moderate, moderately severe, and severe depression respectively

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal Tariq, MSCPPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schilero GJ, Spungen AM, Bauman WA, Radulovic M, Lesser M. Pulmonary function and spinal cord injury. Respir Physiol Neurobiol. 2009 May 15;166(3):129-41. doi: 10.1016/j.resp.2009.04.002. Epub 2009 Apr 9. PMID 19442929
- [Background] Van Houtte S, Vanlandewijck Y, Gosselink R. Respiratory muscle training in persons with spinal cord injury: a systematic review. Respir Med. 2006 Nov;100(11):1886-95. doi: 10.1016/j.rmed.2006.02.029. Epub 2006 Apr 12. PMID 16626951
- [Background] Majdan M, Brazinova A, Mauritz W. Epidemiology of traumatic spinal cord injuries in Austria 2002-2012. Eur Spine J. 2016 Jan;25(1):62-73. doi: 10.1007/s00586-015-3985-z. Epub 2015 May 9. PMID 25957283
- [Background] Darain H, Muhammad Ilyas S, Zeb A, Ullah I, Muhammad D. Epidemiology of Spinal Cord Injury in Pakistan: A Retrospective Study2017. 106-9 p.
- [Background] Roth EJ, Stenson KW, Powley S, Oken J, Primack S, Nussbaum SB, Berkowitz M. Expiratory muscle training in spinal cord injury: a randomized controlled trial. Arch Phys Med Rehabil. 2010 Jun;91(6):857-61. doi: 10.1016/j.apmr.2010.02.012. PMID 20510974
- [Background] Anand S, El-Bashiti N, Sapienza C. Effect of training frequency on maximum expiratory pressure. Am J Speech Lang Pathol. 2012 Nov;21(4):380-6. doi: 10.1044/1058-0360(2012/11-0048). Epub 2012 May 24. PMID 22628108
- [Background] Zupan A, Savrin R, Erjavec T, Kralj A, Karcnik T, Skorjanc T, Benko H, Obreza P. Effects of respiratory muscle training and electrical stimulation of abdominal muscles on respiratory capabilities in tetraplegic patients. Spinal Cord. 1997 Aug;35(8):540-5. doi: 10.1038/sj.sc.3100433. PMID 9267921
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941